CLINICAL TRIAL: NCT05013723
Title: Impact of Monoclonal Antibody Treatment on Post-Acute COVID-19 Syndrome
Acronym: MAbPACs
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: MAbPACs
Record Dates: First submitted 2021-08-02; First posted 2021-08-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Post-acute COVID-19 (PACS), or "long COVID" Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: Patients who received casirivimab-imdevimab antibody infusion
  Interventions: Other: Surveys
- Control: Matched control group who did not receive MAb, matched on diagnosis date, age, gender and Utah COVID-19 Risk Score
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — Mental health validated psychometric surveys: Depression (PHQ-9), Anxiety (GAD-7), PTSD (PC-PTSD-5) Quality of Life surveys: Post COVID-19 Function Status Scale, Quality of life (SF-12)

SUMMARY:
Use the Intermountain real-world MAb-treatment registry and control group to prospectively evaluate PACS symptoms at least 60 days after initial COVID-19 diagnosis.

DETAILED DESCRIPTION:
It is now recognized that many patients who develop symptomatic COVID-19 infection continue to suffer from a variety of symptoms that persist well after the acute syndrome. This has been called post-acute COVID-19 (PACS), or "long COVID" syndrome. In a meta-analysis of studies of hospitalized patients, 70% of patients reported PACS symptoms 60 days after diagnosis. Patients with non-severe COVID-19 appear to have lower rates of PACS symptoms, although a recent study suggested that at 4 months follow-up, 28% of patients still reported at least one symptom. PACS is associated with significant morbidity, decreased quality of life, mental and behavioral health impact and healthcare cost. Neither the pathophysiology nor risk factors for PACS are well-understood and further research is needed to characterize this syndrome. Some studies have suggested that age, female gender, obesity, comorbid burden, symptoms at diagnosis and hospitalization during acute COVID-19 increase risk for PACS. Because of the significant overall impact of PACS, there is significant interest in identifying therapies to prevent this condition. Early neutralizing therapy with anti-SARS-CoV-2 monoclonal antibodies (MAbs) addresses the initial phase of disease and has now been shown to be effective at decreasing viral load and preventing progression to severe disease, hospitalization and death.

Understanding how MAb therapy may impact PACS symptoms is important to determining usage and value of these products and an important contribution to our understanding of how to prevent PACS.

Study Design: Prospective electronic survey using matched case-control design

Objective: Use the Intermountain real-world MAb-treatment registry and control group to prospectively evaluate PACS symptoms at least 60 days after initial COVID-19 diagnosis. Aim 1: Determine whether ambulatory patients who received monoclonal antibody infusion for early symptomatic COVID-19 have fewer persistent symptoms of post-acute COVID-19 ("long COVID") syndrome at least 60 days after initial diagnosis.

Hypothesis: MAb therapy is associated with significantly less post-acute COVID-19 (PACS) symptoms at 120 days post diagnosis Aim 2: Explore predictors associated with PACS symptoms in high risk patients Hypothesis: Hospitalization, age, obesity, number of comorbidities and symptoms at diagnosis predict PACS

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Positive antigen or polymerase chain reaction test for SARS-CoV-2
* Symptomatic COVID-19
* Between day 60 and day 90 from date of positive test
* Not hospitalized or hypoxemic by day 7 of symptoms (Aim 1 only)

Exclusion Criteria:

* Unwilling to participate
* Not able to understand the English language survey questions
* Prisoners
* Inadequate cognitive capacity to provide consent and complete the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with laboratory-confirmed acute COVID-19 in the Intermountain MAb registry, assessed at least 60 after positive test date but no greater than 90 days
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Post-acute COVID-19 symptom score (out of 60) | Between day 60 and day 90 from date of positive test
  Post-acute COVID-19 symptom score (out of 60)

SECONDARY OUTCOMES:
Medically attended visits | Between day 60 and day 90 from date of positive test
  Number of medically attended visits between day 60 and day 90 from date of positive test
Healthcare costs | Between day 60 and day 90 from date of positive test
  Total healthcare costs to health system
Diagnostic test costs | Between day 60 and day 90 from date of positive test
  Total diagnostic test costs to health system
Mental health validated psychometric surveys: Depression (PHQ-9),PTSD (PC-PTSD-5) | Between day 60 and day 19 from date of positive test
  Depression (PHQ-9) score. Range (0-27). Lower scores indicate better health
Post COVID-19 Function Status Scale | Between day 60 and day 90 from date of positive test
  Quality of Life surveys: Post COVID-19 Function Status Scale. Range (0-4), lower score indicates better health
Mental health validated psychometric survey: Anxiety (GAD-7) | Between day 60 and day 90 from date of positive test
  Anxiety (GAD-7) score (Range 0 -21). Lower scores indicate better health
Quality of life (SF-12) | Between day 60 and day 90 from date of positive test
  SF-12 Short Form 12. Range (0-64), high scores indicate better health
Primary Care Post-Traumatic Stress Disorder 5 | Between day 60 and day 90 from date of positive test
  PTSD-5. Range (0-5); lower scores indicate better health

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No